CLINICAL TRIAL: NCT07187999
Title: Dental Morphometric Correlation Between Crown Dimensions to Physical Height of a Child
Brief Title: Dimensional Correlation Between Tooth Measurements and Physical Height in Children
Status: Completed | Type: Observational
Sponsor: Rungta College of Dental Sciences and Research (Other)
Responsible Party: Principal Investigator, Karthik Krishna M, Professor, Rungta College of Dental Sciences and Research
Other Study IDs: RCDSR/IEC/MDS/2023/D15
Record Dates: First submitted 2025-09-08; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-03

CONDITIONS: Relationship Between the Physical Height and the Clinical Crown Length in Children
Keywords: growth retardation; stature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children of 3-6 years age

SUMMARY:
Correlation between height of a child and their teeth dimensions needs to be established for several reasons such as determination of growth of an individual (growth records), growth spurts and medicolegal issues. This study was performed to evaluate this relationship.

DETAILED DESCRIPTION:
A total of 210 samples of deciduous dentition from children aged 3-6 years were collected. Impressions were taken using elastomeric material, and casts were created with Type IV die stone. A digital vernier caliper measured the clinical crown length, which was correlated with the child's physical height.

Statistical analysis revealed significant correlations between certain primary teeth and height in children. Based on the findings, mathematical equations were developed to predict physical height based on crown length.

ELIGIBILITY:
Inclusion Criteria:

* Age: 3-6 years old
* Fully erupted maxillary and mandibular right quadrant teeth.
* Healthy state of gingiva and periodontium.
* No crowding or malpositioned teeth.

Exclusion Criteria:

* Loss of tooth structure due to fracture, attrition, or dental caries may impact study results
* Children with congenital dental anomalies or systemic conditions affecting oral health
* Previous dental treatment or restoration
* Special needs or behavioral issues

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 210 children who met the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Physical Height | Baseline
Crown height | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatric Dentistry, Rungta College of Dental Sciences and Research, Bhilai, Chhattisgarh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sruthi R, Reddy RS, Rajesh N, Jyothirmai K, Preethi M, Teja TN. Carrea's Index and Tooth Dimensions- An Avant-Garde in Stature Estimation: An Observational Study. J Clin Diagn Res. 2016 Dec;10(12):ZC33-ZC37. doi: 10.7860/JCDR/2016/22646.9046. Epub 2016 Dec 1. PMID 28209000
- [Background] FILIPSSON R, GOLDSON L. CORRELATION BETWEEN TOOTH WIDTH, WIDTH OF THE HEAD, LENGTH OF THE HEAD, AND STATURE. Acta Odontol Scand. 1963 Nov;21:359-65. doi: 10.3109/00016356309028200. No abstract available. PMID 14110645